CLINICAL TRIAL: NCT01346813
Title: Epidémiologie Des Gestes Douloureux ou Stressants Chez Les Nouveau-nés Pris en Charge Dans Les unités de réanimation néonatale et pédiatrique et Par Les équipes de SMUR de la région d'Ile de France
Brief Title: Epidemiology of Painful Procedures in Neonates
Acronym: EPIPPAIN
Status: Completed | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, CARBAJAL, Professor, Hôpital Armand Trousseau
Other Study IDs: EPIPPAIN2_IDF
Record Dates: First submitted 2011-05-02; First posted 2011-05-03 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Newborn Morbidity; Pain; Procedures; Intratracheal Intubation; Analgesia; Intensive Care; Longterm Effects
Keywords: Newborns; Premature; Pain; Pain assessment; Painful Procedures; Stressful Procedures; Endotracheal Intubation; Analgesia; Sedation; Longterm effects of pain; Epidemiology
MeSH Terms: conditions — Pain; Agnosia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sick or premature neonates are exposed to frequent painful and stressful procedures during their stay in neonatal intensive care units. Although neonates do feel pain and may have long term effects induced by painful experiences, prevention and treatment of neonatal pain is far from optimal in many units. An epidemiological study (EPIPPAIN) conducted in neonatal and pediatric intensive care units in France in 2005 showed that painful procedures were extremely frequent and that analgesics treatments varied a lot among units. Since many guidelines have been issued by international scientific societies to manage neonatal pain, one may expect that the prevention and treatment of neonatal pain has improved over the last 6 years.

Although awake endotracheal intubations are extremely difficult or impossible in older children or adults, such intubations are still frequently performed without sedation/analgesia in neonates. Recent studies have shown that premedications facilitate intubation conditions and greatly improve neonates tolerance of the procedure. Studies aimed at assessing the risks and benefits of different sedations/analgesia strategies are urgently needed in neonates. We also need a tool to assess at the same time the technical conditions of intubations and the tolerance of the neonate to the procedure so that data from different studies can be compared.

The objectives of the present study are:

1. To describe the incidence of painful and stressful procedures performed in the neonate in intensive care units as well as in neonates transported by the medical emergency system (SMUR) of the Ile-de-France region 6 years after the first EPPIPAIN study conducted in the same region and same type of population in order to assess the evolution of practices. The description of painful and stressful procedures will be completed with a real-time around-the-clock assessment of the pain induced by procedures using a validated behavioral pain scale.
2. To link this study with The Epipage study 2 in order to look for associations between the number of painful and stressful procedures and/or analgesic treatments of the neonatal period and the neurological outcome of children that will be followed in the Epipage cohort. The Epipage study is a separate study that will follow for 13 years a cohort of premature neonates recruited in 2011.
3. To describe the incidence of painful or stressful procedures and analgesic treatments in neonates transported by the pediatric emergency system (SMUR) of the Ile-de-France region in France.
4. To obtain initial validity of a tool permitting to assess intubations in neonates. An observational detailed description of endotracheal intubations conditions will be conducted in neonates transported and intubated by SMUR and in neonates intubated in intensive care units
5. To describe continuous sedation and analgesia practices in ventilated neonates in intensive care units. For these neonates, data from medical records will be recovered up to 2 months of admission in intensive care units
6. To describe the frequency of heel sticks for glycemia measurement and blood gazes practices among centers. Relate heel stick practices to the normality or abnormality of glycemia results

DETAILED DESCRIPTION:
STUDY HYPOTHESIS

Principal hypothesis

- The number of painful and stressful procedures performed in the neonate admitted to intensive care units is still very high but it is lower than in 2005 Pain scores are lower when procedures are performed with a specific analgesia prior to procedure.

Secondary hypothesis

* The frequency of pre-procedural analgesia is higher than in 2005
* Certain common procedures such as heel sticks and endotracheal intubations are carried out with a more frequent analgesia than in 2005
* The use of a continuous sedation and analgesia does not induce a reduction in specific pre-procedural analgesia
* A real-time pain assessment of painful procedures can be carried out in more than 80% of procedures performed in neonates in intensive care units Pain scores show that certain procedures which are apparently not very painful may elicit high pain scores in very sick neonates
* Certain procedures such as nursing care or weighing may induce high pain scores in neonates who have invasive tubes (endotracheal tubes, thoracic drainage)
* A continuous sedation and analgesia is given to more than 50% of ventilated neonates.
* Certain characteristics of neonates may influence the use of analgesics for painful procedures. Ex: gender, age, respiratory support
* Certain contextual characteristics or center may influence the use of analgesics for painful procedures. Ex: day or night, pain referent in the unit, night head nurse, written pain management guidelines.
* More than 80% of semi-urgent or non-urgent intubations are carried out with the use of premedication.
* Opioids are the most commonly drugs used for premedication during endotracheal intubations in neonates
* The assessment of intubating conditions and neonate tolerance show lower scores when intubations are performed with a premedication considered as "recommended" by the American Academy of Pediatrics
* The detailed observation of intubations in SMUR and intensive care units will enable initial validation of a tool assessment
* Too many capillary blood samples by heel sticks are carried out in neonates even in neonates that have normal values throughout repeated sticks.
* The frequency of blood gas assessments is widely variable among centers
* The frequency of capillary blood glycemia is widely variable among centers

LONG-TERM EFFECTS OF PAIN AND ANALGESIC TREATMENTS

This objective will be assessed by matching the data of the current Epippain study and another parallel study (Epipage 2)

Principal hypothesis

- After adjusting for the disease severity, neonates that undergo more painful procedures have a poorer neurological outcome later in infancy.

Secondary hypothesis

* Higher pain scores are associated with a poorer neurological outcome later in infancy
* The use of central analgesics like opioid does not have a negative effect on neurological outcome later in infancy.
* The potential negative effect of numerous painful procedures during the neonatal period can be counteracted by the use of analgesics.

METHODOLOGY

This study will be carried out in neonates cared for in two settings: (i) neonatal or pediatric intensive care units and (ii) the medical regional pediatric transport system (SMUR) In the intensive care units, this study is designed as a prospective observational study to collect around-the-clock bedside data on all painful or stressful procedures performed in neonates admitted to the participating units. All 16 tertiary care centers, Neonatal Intensive Care Units (NICUs) and Pediatric Intensive Care Units (PICUs) in the Paris Region will participate. Since this is an observational study no changes in the standard of care will be carried out. During the first 14 days of admission to the participating units, prospective data will be collected on all neonatal procedures causing pain, stress, or discomfort with the corresponding analgesic therapy. A real-time assessment of pain induced by each procedure will be carried out by unit staff using the DAN scale. A detailed record of conditions of endotracheal intubations will also be carried out.

Demographic data, type and duration of respiratory support, sedative and analgesic drugs administered concomitantly or pre-procedure, and conditions related to each procedure (type, hour of the day, operator, parental presence) will be collected. We'll also record repeat procedure attempts for procedures requiring more than one attempt before successful completion. The use of specific pre-procedural analgesia will be noted for each procedure. If neonates are discharged from the units before 14 days, data collection on painful procedures will be stopped on the day of discharge.

In the medical regional pediatric transport system (SMUR), neonates transported during the 2-months study period, will have all their procedures recorded in a specific data collection form. Demographic data, type of respiratory support, sedative and analgesic drugs administered concomitantly or pre-procedure, and conditions related to each procedure (type, hour of the day, operator, parental presence) will be collected. We'll also record repeat procedure attempts for procedures requiring more than one attempt before successful completion. The use of specific pre-procedural analgesia will be noted for each procedure. A real-time assessment of pain induced by each procedure will be carried out by unit staff using the DAN scale. A detailed record of conditions and neonate tolerance of endotracheal intubations will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

Intensive care units:

* Neonates admitted to the unit during the 6-week recruitment period
* Age less than 45 post-conceptional weeks

Regional pediatric transport system (SMUR):

* Neonates transported during the 2-months recruitment period
* Age less than 45 post-conceptional weeks

Exclusion Criteria:

* None

Max Age: 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Two settings: neonatal or pediatric intensive care units and regional pediatric transport system (SMUR).
  In intensive care units, during the first 14 days of admission prospective data will be collected on all neonatal procedures causing pain, stress, or discomfort with the corresponding analgesic therapy and pain assessment. A detailed record of conditions of endotracheal intubations will also be carried out.
  In the SMUR, neonates transported during the 2-months study period by all of 5 SMUR will have all their procedures recorded in a specific data collection form. A real-time assessment of pain induced by each procedure will be carried out by staff using the DAN scale. A detailed record of conditions and neonate tolerance of endotracheal intubations will also be carried out.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Carbajal, MD, PhD, Principal Investigator — Hôpital Armand Trousseau, Paris, France
Locations (21):
- France (21):
  - Hôpital Victor Dupouy. Service de réanimation néonatale, Argenteuil
  - Hôpital Antoine Béclère. Service de réanimation néonatale, Clamart
  - SMUR 92 Clamart, Clamart
  - Hôpital Louis Mourier. Service de réanimation néonatale, Colombes
  - CHI Créteil. Service de réanimation néonatale, Créteil
  - Hôpital du Sud Francilien. Service de réanimation néonatale, Évry
  - Hôpital de Bicêtre. Service de réanimation pédiatrique et néonatale, Le Kremlin-Bicêtre
  - Hôpital de Meaux. Service de réanimation néonatale, Meaux
  - CHI André Grégoire. Service de réanimation néonatale, Montreuil
  - SAMU 93 Montreuil, Montreuil
  - Hôpital Armand Trousseau. Service de Réanimation Pédiatrique, Paris
  - Hôpital Cochin-Port Royal. Service de médecine néonatale, Paris
  - Institut de Puériculture et de Périnatalogie. Service de réanimation néonatale, Paris
  - Hôpital Necker Enfants Malades. Service de réanimation pédiatrique et néonatale, Paris
  - SMUR 75 Necker, Paris
  - Hôpital Robert Debré. Service de réanimation néonatale, Paris
  - SMUR 75 Robert Debré, Paris
  - Centre Hospitalier Intercommunal de Poissy Saint Germain en Laye Service de réanimation néonatale, Poissy
  - Centre Hospitalier René Dubos. Service de réanimation néonatale, Pontoise
  - SAMU 95 Pontoise, Pontoise
  - Hôpital Delafontaine. Service de réanimation néonatale, Saint-Denis

REFERENCES:
- [Derived] Carbajal R, Lode N, Ayachi A, Chouakri O, Henry-Larzul V, Kessous K, Normand A, Courtois E, Rousseau J, Cimerman P, Chabernaud JL. Premedication practices for tracheal intubation in neonates transported by French medical transport teams: a prospective observational study. BMJ Open. 2019 Nov 14;9(11):e034052. doi: 10.1136/bmjopen-2019-034052. PMID 31727669
- [Derived] Courtois E, Cimerman P, Dubuche V, Goiset MF, Orfevre C, Lagarde A, Sgaggero B, Guiot C, Goussot M, Huraux E, Nanquette MC, Butel C, Ferreira AM, Lacoste S, Sejourne S, Jolly V, Lajoie G, Maillard V, Guedj R, Chappuy H, Carbajal R. The burden of venipuncture pain in neonatal intensive care units: EPIPPAIN 2, a prospective observational study. Int J Nurs Stud. 2016 May;57:48-59. doi: 10.1016/j.ijnurstu.2016.01.014. Epub 2016 Feb 8. PMID 27045564